CLINICAL TRIAL: NCT03049267
Title: Short-term Safety, Efficacy and Mode of Action of Apremilast in Moderate Suppurative Hidradenitis: A Randomised Double-blind Placebo Controlled Trial
Brief Title: Short-term Safety, Efficacy and Mode of Action of Apremilast in Moderate Suppurative Hidradenitis
Acronym: SMASH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.B.A. van Doorn (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor-Investigator, M.B.A. van Doorn, MD, PhD, Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SMASH trial
Record Dates: First submitted 2016-10-25; First posted 2017-02-10 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Hidradenitis Suppurativa
Keywords: acne inversa
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — apremilast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Apremilast (Experimental): N=15
  Interventions: Drug: Apremilast
- Placebo Oral Tablet (Placebo Comparator): N=5
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Apremilast — Fifteen patients will be supplied of apremilast for daily oral use; 16 weeks.
  Other Names: Otezla, CC-10004
  Arms: Apremilast
Drug: Placebo Oral Tablet — Five patients will be supplied with placebo tablets with identical labeling as apremilast for daily use; 16 weeks.
  Other Names: Placebo comparator
  Arms: Placebo Oral Tablet

SUMMARY:
Study design: A double-blind randomised placebo-controlled trial

Intervention: Randomized placebo controlled treatment of 20 HS patients of which fifteen patients will be randomized to apremilast and five patients to placebo. The total duration of the treatment period per subject is 16 weeks.

Primary objectives: To evaluate the expression profile of inflammatory cytokines in HS lesional skin at week four (t=4) and week sixteen (t=16):

* of patients receiving apremilast compared to placebo;
* within both groups relative to baseline (t=0).

Secondary objectives:

* To prospectively evaluate the clinical efficacy of apremilast.
* To assess the effect of apremilast on patient reported outcomes measures.
* To assess the short-term safety and tolerability of apremilast in patients with hidradenitis suppurativa.

DETAILED DESCRIPTION:
Rationale:

Hidradenitis suppurativa (HS) is a chronic, inflammatory, recurrent, debilitating skin disease. It is characterized by painful, deep-seated, inflamed boils in the inverse areas of the body, most commonly the axillae, inguinal and anogenital regions.

Systemic therapy with immunosuppressive agents (systemic corticosteroids, dapsone, cyclosporin) has been investigated in the past decades and has shown limited efficacy. The use of the selective immunosuppressant apremilast has not yet been evaluated in HS. The investigators hypothesize a beneficial effect of apremilast in HS patients, similar to the efficacy of apremilast in psoriasis patients. Namely, it has been shown that the immune dysregulation in the pathogenesis of HS shows many similarities with that of psoriasis. Moreover, the TNF-α blocker adalimumab was registered for HS after approval for the treatment in patients with psoriasis.

ELIGIBILITY:
Key inclusion criteria:

* Adult (≥ 18 years of age) male or female patients with moderate HS according to a PGA of 3 on the 5-point HS-Physician Global Assessment (HS-PGA);
* HS of more than 6 months duration; have lesions in at least two anatomical locations.

Key exclusion criteria:

* Contra-indication for apremilast; previous use of apremilast; have any current and/or recurrent clinically significant skin condition in the treatment area other than HS;
* Presence of other uncontrolled major disease;
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2017-12-06 (Actual); Study Completion 2018-06-28 (Actual)

PRIMARY OUTCOMES:
Change of expression levels of inflammatory cytokine mRNA in HS lesional skin. | t=16 weeks
  measurement by qPCR
Change of expression levels of inflammatory cytokine protein in HS lesional skin. | t=16 weeks
  measurement by ELISA

SECONDARY OUTCOMES:
Abscesses count | t=0 weeks, t=4 weeks, t=16 weeks
  Total number of abscesses [A]
Nodule count | t=0 weeks, t=4 weeks, t=16 weeks
  Total number of inflammatory [N] and non-inflammatory nodules
Fistula count | t=0 weeks, t=4 weeks, t=16 weeks
  Total count of draining fistulas
Hidradenitis Suppurativa Physician's Global Assessment (HS-PGA) score | t=0 weeks, t=4 weeks, t=16 weeks
  Based on the HS lesion count
Hidradenitis Suppurativa Clinical Response (HiSCR) | t=0 weeks, t=16 weeks
  Based on the AN count; The proposed definition of 50% and 30% responders to treatment (HiSCR achievers) is respectively: (i) at least a 50% and 30% reduction in ANs, (ii) no increase in the number of abscesses, and (iii) no increase in the number of draining fistulas from baseline.
Numerical Rating Scale (NRS) | t=0 weeks, t=4 weeks, t=16 weeks
  To assess the patient reported outcome measures (PROMs) pain, pruritus and patient disease global assessment score;
Dermatology Life Quality Index (DLQI) | t=0 weeks, t=4 weeks, t=16 weeks
  To assess the patient reported outcome measures (PROM) quality of life
Incidence of Treatment-Emergent Adverse Events | Multiple time points between t=0 weeks and t=16 weeks
  Vital signs: heart rate, temperature, blood pressure. Patient reported adverse events Safety laboratories: White blood cell count, Absolute neutrophil count, Hemoglobin, Platelets, Serum Creatinine, ALT, Alkaline phosphatase

CONTACTS AND LOCATIONS:
Overall Officials: Errol Prens, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus University Medical Center, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No